CLINICAL TRIAL: NCT01691079
Title: Effectiveness of Ipratropium Bromide in Preventing Exercise-induced Bronchoconstriction in Athletes
Acronym: STAMINA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-09621
Record Dates: First submitted 2012-09-13; First posted 2012-09-24 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Bronchospasm, Exercise-Induced
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — Ipratropium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): placebo 2 puffs prior to exercise challenge
  Interventions: Drug: Placebo
- ipratropium bromide (Active Comparator): ipratropium bromide HFA 2 puffs prior to exercise challenge
  Interventions: Drug: ipratropium bromide

INTERVENTIONS:
Drug: ipratropium bromide — Inhaled ipratropium bromide administered before exercise.
  Other Names: atrovent
  Arms: ipratropium bromide
Drug: Placebo — Inhaled placebo administered before exercise.
  Arms: placebo

SUMMARY:
This will be a double-blind placebo-controlled study in which we plan to study 40 competitive endurance athletes. We will conduct an exercise test to evaluate maximal oxygen uptake and 2 exercise challenge tests to provoke EIA. Prior to the exercise challenge tests the athletes will randomly receive inhaled placebo or inhaled ipratropium bromide. We will compare the athletes' airway response to the exercise challenge with and without the active drug.

DETAILED DESCRIPTION:
Exercise-induced asthma (EIA) is common and often unrecognized among endurance athletes. The mechanisms of asthma appear to be different between athletes and non-athletes, in that the occurrence of asthma is higher among endurance athletes and seems to be promoted by training. This suggests that factors inherent to athleticism, such as the parasympathetic nervous system, which has been shown to change with endurance training and is known to lead to narrowing of the airways, may be involved with the development of asthma in athletes. Although asthma mechanisms and treatments have been extensively studied in classic asthmatics, there is very limited data in athletes.

This will be a double-blind placebo-controlled study in which we plan to study 40 competitive endurance athletes. We will conduct an exercise test to evaluate maximal oxygen uptake and 2 exercise challenge tests to provoke EIA. Prior to the exercise challenge tests the athletes will randomly receive inhaled placebo or inhaled ipratropium bromide. We will compare the athletes' airway response to the exercise challenge with and without the active drug.

If ipratropium bromide proves to prevent EIA in athletes, this drug may be appropriate and effective to target EIA in this population. The results of this study may lead to improved clinical management of athletes with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Athletes > 13 years of age

Exclusion Criteria:

* History of cardiac complaints (chest pain, shortness of breath, palpitations, dyspnea on exertion).
* History of cardiac disease or taking cardioactive medications.
* History of smoking.
* History of glaucoma.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mona Luke-Zeitoun, Principal Investigator — Assistant Clinical Professor (Volunteer)
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PI left institution and sincere efforts were made to contact the PI, but were unsuccessful. No data are available to report.
Period: Overall Study
Arm/Group | Placebo | Ipratropium Bromide
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: PI left institution and sincere efforts were made to contact the PI, but were unsuccessful. No data are available to report.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ipratropium Bromide | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Spirometry and Specific Airway Conductance Measured by Body Plethysmography Before and After Exercise Challenge After Randomized Administration of Either Inhaled Ipratropium Bromide or Inhaled Placebo
Time Frame: The outcome measures will be assessed over an expected average of 6 months.
Population: as for baseline characteristics
Arm/Group | Placebo | Ipratropium Bromide
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Specific IgE Measurements
Time Frame: The outcome measures will be assessed over an expected average of 6 months.
Population: as for baseline characteristics
Arm/Group | Placebo | Ipratropium Bromide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: PI left institution and sincere efforts were made to contact the PI, but were unsuccessful. No data are available to report.
Arm/Group | Placebo | Ipratropium Bromide
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes